CLINICAL TRIAL: NCT07136649
Title: Effects of Custom CAD/CAM Insoles on Plantar Pressure Distribution in Individuals With Foot Deformities: A Randomized Controlled Trial
Brief Title: Custom CAD/CAM Insoles for Plantar Pressure Improvement in Foot Deformities
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Başar Öztürk, Associate Professor, Department of Physiotherapy and Rehabilitation (English), Faculty of Health Sciences, Fenerbahçe University, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: assoc.prof.basarozturk
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Foot Deformities; Orthotic Device; 3D Printing; CAD
Keywords: Custom CAD/CAM Insoles; Pes Planus; Pes Planovalgus; Pes Cavus; Pedobarography; Plantar Pressure; 3D Printing; Orthotics
MeSH Terms: conditions — Foot Deformities; Flatfoot; Clubfoot; Talipes Cavus

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the intervention group, receiving custom CAD/CAM insoles, or the control group, receiving no insole intervention, with both groups assessed at baseline and after eight weeks.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to group allocation to prevent measurement bias during data collection and analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Custom CAD/CAM Insole Group (Experimental): Participants in this group will receive custom CAD/CAM insoles designed based on 3D plantar scans and pedobarographic analysis. The insoles will be fitted into their regular footwear and used daily for eight consecutive weeks.
  Interventions: Device: Custom CAD/CAM Insoles
- Control Group (No Insole Intervention) (No Intervention): Participants in this group will not receive any insole intervention during the eight-week study period and will continue using their usual footwear.

INTERVENTIONS:
Device: Custom CAD/CAM Insoles — Custom insoles will be designed using 3D plantar scanning and pedobarographic analysis, produced with CAD/CAM technology. The insoles will be fitted into participants' regular footwear and worn daily for eight consecutive weeks. The design aims to optimize plantar pressure distribution and improve foot biomechanics in individuals with foot deformities.
  Arms: Custom CAD/CAM Insole Group

SUMMARY:
This randomized controlled trial will investigate the effects of custom CAD/CAM insoles on plantar pressure distribution and gait parameters in individuals with foot deformities, such as pes planus, pes cavus, and hallux valgus. A total of 30 participants will be randomly assigned to either the intervention group, receiving custom CAD/CAM insoles, or the control group, receiving no insole intervention.

Plantar pressure measurements will be performed using the As200 Gait Scan Pedobarography System at baseline and after eight weeks. Static and dynamic plantar pressure variables, contact area, and center of pressure displacement will be assessed, along with gait parameters including step length, step time, and walking speed.

The results of this study may contribute to the development of effective conservative treatment strategies to improve foot biomechanics and reduce pressure-related complications in individuals with foot deformities.

DETAILED DESCRIPTION:
This randomized controlled trial will evaluate the impact of custom CAD/CAM insoles on plantar pressure distribution and gait parameters in individuals with clinically diagnosed foot deformities. Thirty eligible participants, aged 18-65 years, will be randomly assigned to one of two groups:

Intervention Group: Participants will receive custom-designed CAD/CAM insoles based on 3D plantar scans and pedobarographic analysis.

Control Group: Participants will not receive insole intervention during the eight-week study period.

Baseline assessments will include demographic data, anthropometric foot measurements, and pedobarographic analysis using the As200 Gait Scan System. The intervention group will be instructed to use the custom insoles daily for eight consecutive weeks, while the control group will maintain their usual footwear without insoles.

After eight weeks, all participants will undergo the same measurement procedures. Primary outcome measures will include maximum and mean plantar pressures, contact area, and center of pressure displacement. Secondary outcomes will include step length, step time, walking speed, and regional pressure distribution across foot segments.

Data analysis will be conducted using repeated-measures statistical models to evaluate time × group effects, with significance set at p < 0.05. The study will be conducted at the Kale Prosthetics and Orthotics Center between September and November 2025, following approval from the Fenerbahçe University Non-Interventional Clinical Research Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* Clinically diagnosed with a foot deformity (e.g., pes planus, pes cavus, hallux valgus)
* Able to use custom insoles for at least six months
* Able to stand and walk for pedobarographic measurements
* Willing to participate and provide informed consent

Exclusion Criteria:

* Presence of neurological or systemic diseases affecting foot function (e.g., diabetic neuropathy)
* History of lower extremity surgery in the last six months
* Severe musculoskeletal conditions impairing sensorimotor function
* Any condition preventing compliance with insole use
* Contraindications for participating in gait or pressure measurements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Plantar Pressure | Baseline and 8 weeks after intervention.
  Maximum plantar pressure (kPa) measured under static and dynamic conditions using the As200 Gait Scan Pedobarography System.
Mean Plantar Pressure | Baseline and 8 weeks after intervention.
  Mean plantar pressure (kPa) measured under static and dynamic conditions using the As200 Gait Scan Pedobarography System.
Plantar Contact Area | Baseline and 8 weeks after intervention.
  Plantar contact area (cm²) measured under static and dynamic conditions using the As200 Gait Scan Pedobarography System.
Center of Pressure (COP) Displacement | Baseline and 8 weeks after intervention.
  Center of pressure (COP) displacement (mm) measured under static and dynamic conditions using the As200 Gait Scan Pedobarography System.

SECONDARY OUTCOMES:
Step Length | Baseline and 8 weeks after intervention
  Step length (cm) assessed using the As200 Gait Scan Pedobarography System under dynamic walking conditions.
Step Time | Baseline and 8 weeks after intervention
  Step time (ms) assessed using the As200 Gait Scan Pedobarography System under dynamic walking conditions.
Walking Speed | Baseline and 8 weeks after intervention.
  Walking speed (m/s) assessed using the As200 Gait Scan Pedobarography System under dynamic walking conditions.
Regional Pressure Distribution | Baseline and 8 weeks after intervention.
  Plantar pressure distribution by foot regions (kPa) assessed using the As200 Gait Scan Pedobarography System.

OTHER OUTCOMES:
Arch Height | Baseline and 8 weeks after intervention.
  Arch height (cm) measured using a digital caliper and measuring tape.
Navicular Drop | Baseline and 8 weeks after intervention.
  Navicular drop (mm) measured using a digital caliper and measuring tape.
Hallux Valgus Angle | Baseline and 8 weeks after intervention.
  Hallux valgus angle (degrees) measured using a goniometer.

IPD SHARING:
Plan to Share IPD: No